CLINICAL TRIAL: NCT04486066
Title: An Evaluation of MBSR and CBT for Veterans With Chronic Pain
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3283-R; IO1RX003283-01A2 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Pain
Keywords: mindfulness; cognitive behavioral therapy
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Mindfulness-Based Stress Reduction; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): In MBSR, participants meet for 2 hours per week for 8 weeks in a video group format and receive instruction in mindfulness meditation according to a standardized curriculum, are given daily homework, participate in group discussions, and can ask questions.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) (Experimental): Cognitive Behavioral Therapy (CBT) is the most widely used non-pharmacologic intervention for chronic pain and a version of CBT specifically addressing chronic pain (CBT-CP) has been developed for use in VA with Veterans. Fundamentally, CBT is an approach that seeks to ameliorate dysfunctional relationships between an individual's thoughts, feelings, and behaviors to improve functioning and quality of life. At our site, the CBT-CP format has been adapted for clinical use (i.e., as part of usual clinical care) to 8 sessions in a video group format, while retaining all essential elements.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain
- Usual Care (Other): Veterans randomized to usual care will continue to be followed by their usual care providers for all medical and mental health care. This can include continued use of medications, specialty referrals and other usual elements of care. They will be asked to not enroll in the specific MBSR or CBT-CP interventions during the 8-month study period, but can attend other groups interventions, such as CBT-Insomnia, Acceptance and Commitment Therapy for Chronic Pain, and other groups for chronic pain and PTSD as directed by their treating providers. They can also enroll in MBSR or CBT-CP at the completion of the study.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — In MBSR, participants meet by video for 2 hours per week for 8 weeks in a group format and receive instruction in mindfulness meditation according to a standardized curriculum, are given daily homework, participate in group discussions, and can ask questions.
  Arms: Mindfulness-Based Stress Reduction (MBSR)
Behavioral: Cognitive Behavioral Therapy for Chronic Pain — Cognitive Behavioral Therapy (CBT) is the most widely used non-pharmacologic intervention for chronic pain and a version of CBT specifically addressing chronic pain (CBT-CP) has been developed for use in VA with Veterans. Fundamentally, CBT is an approach that seeks to ameliorate dysfunctional relationships between an individual's thoughts, feelings, and behaviors to improve functioning and quality of life. At our site, the CBT-CP format has been adapted for clinical use (i.e., as part of usual clinical care) to 8 video sessions in a group format, while retaining all essential elements.
  Arms: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)
Other: Usual Care — Veterans randomized to usual care will continue to be followed by their usual care providers for all medical and mental health care. This can include continued use of medications, specialty referrals and other usual elements of care. They will be asked to not enroll in the specific MBSR or CBT-CP interventions during the 8-month study period, but can attend other groups interventions, such as CBT-Insomnia, Acceptance and Commitment Therapy for Chronic Pain, and other groups for chronic pain and PTSD as directed by their treating providers. They can also enroll in MBSR or CBT-CP at the completion of the study.
  Arms: Usual Care

SUMMARY:
Approximately fifty percent of Veterans report chronic pain. Management of chronic pain is often compounded by other life problems, including depression and posttraumatic stress disorder. Use of opioids for pain management entails risk of harm, and effective non-pharmacologic approaches to chronic pain management are needed. Mindfulness-Based Stress Reduction (MBSR) and group Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) are programs that teach skills to improve functionality and quality of life for people with chronic pain. However, studies of MBSR and the group form of CBT-CP for chronic pain remain limited. In the proposed trial, MBSR will be compared to CBT-CP and usual care, with assessment of pain interference and other outcomes at 6-month follow-up. If MBSR and group CBT-CP are shown to be effective in improving outcomes, it would support use of these modalities for chronic pain.

DETAILED DESCRIPTION:
Background: Pain is one of the most common reasons Veterans seek health care. Mental health conditions (including PTSD, anxiety, and depression) are estimated to co-occur for 30-50% of Veterans with chronic pain. Current recommendations for pain management include an integrative approach informed by the biopsychosocial model. It is increasingly recognized that use of opioids for pain management is associated with risk of harm, yet treatment studies of non-pharmacologic approaches remain limited. Mindfulness-Based Stress Reduction (MBSR) and Cognitive Behavioral Therapy for chronic pain (CBT-CP) teach skills intended to enhance functionality and quality of life in the face of chronic pain. The proposed randomized clinical trial will evaluate if MBSR and CBT-CP each result in improvements in pain interference that are superior to usual care. Two hundred twenty-two Veterans with chronic musculoskeletal pain will be randomized to MBSR, CBT-CP or usual care. Measures pertaining to the primary outcome of pain interference will be collected at baseline, at the post-MBSR/CBT-CP time point, and at 6-month follow-up. In addition, measures of pain intensity, depression, and treatment satisfaction will be applied to more fully characterize the impact of MBSR relative to CBT-CP and usual care. Exploratory analyses will assess if outcomes differ for MBSR and CBT-CP, the impact of the interventions on opioid use and indicators of suicidality, and whether Veteran characteristics assessed at baseline function as treatment moderators. Aims: Primary Aim: Assess if MBSR and CBT-CP each result in greater reductions in the pain interference subscale of the Brief Pain Inventory (BPI) as compared to usual care, from baseline to 6 months post-treatment. Secondary Aim: Evaluate if MBSR and CBT-CP are each superior to usual care in producing improvements in pain severity, treatment satisfaction, and depression. Exploratory Aim 1: Evaluate whether outcomes for patients randomized to MBSR and CBT-CP differ for changes in pain interference, pain severity, depression, and treatment satisfaction. Exploratory Aim 2: Evaluate the impact of MBSR and CBT-CP on utilization of opioid analgesics and markers of suicidality.

Exploratory Aim 3: Evaluate moderators of response to MBSR and CBT-CP to lay the groundwork for identifying Veterans more likely to succeed in one or the other treatment. Potential moderators assessed will include: age, gender, baseline depressive symptoms, anxiety sensitivity, and pain catastrophizing.

Design: A three-arm randomized controlled trial comparing MBSR, CBT-CP and usual care. Participants: 222 Veterans at a large urban VA facility with chronic musculoskeletal pain. Interventions: Group MBSR or group CBT-CP, each 8 weeks in duration. Analyses: Mixed models with assess whether MBSR, CBT-CP each produce greater reductions in outcome variables from baseline to follow-up compared to usual care. Implications: If MBSR and CBT-CP are each shown to be superior to usual care for treatment of chronic pain among Veterans, it would support providing MBSR and CBT-CP for this population.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet criteria for chronic musculoskeletal pain, defined as:

* musculoskeletal pain of low back
* cervical spine, or extremities (hip, knee, or shoulder)
* pain for at least 3 months
* pain severity (worst or average pain score equal to or greater than 4)(i.e., score of 4 or greater on BPI items 3 or 5) and average pain interference (BPI items 9A-9G) rated equal to or great than 3 of 10 over prior week, as measured using the Brief Pain Inventory (BPI)

Exclusion Criteria:

At baseline, the MINI psychiatric interview will determine psychiatric exclusion criteria:

* uncontrolled psychotic disorder
* current bipolar affective disorder with mania
* current suicidal or homicidal ideation with intent in the last month
* inpatient psychiatric admission within the past month
* severe medical conditions that would limit participation (e.g., Class III or IV heart failure)
* pending back surgery

Additional exclusion criteria include prior formal participation in MBSR or CBT-CP. The investigators will include subjects with Alcohol Use Disorder (AUD; defined by the MINI) but exclude those for whom alcohol use poses a safety threat (defined as current drinking and a past-year history of alcohol-related seizures or delirium tremens). The investigators will also include those with Opioid Use Disorder (OUD) and other Substance Use Disorder (SUD; each defined by the MINI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Simpson, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction (MBSR) | Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) | Usual Care
Started (Number randomized to each condition.) | 75 | 71 | 71
Completed Treatment (Completed intervention (attended 6 of 8 sessions)) | 48 | 55 | 0 (The usual care condition did not have set appointments so there was no "treatment completion" metric.)
Post-treatment Assessment | 68 | 68 | 70
Completed (Completed final 6-month assessment) | 66 | 65 | 69
Not Completed | 9 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction (MBSR) | Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) | Usual Care | Total
Number analyzed (Participants) | 75 | 71 | 71 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 40 | 116
  >=65 years | 37 | 33 | 31 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.9) | 60.8 (13.9) | 61.0 (12.6) | 61.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 13 | 40
  Male | 60 | 59 | 58 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 11 | 4 | 18
  Not Hispanic or Latino | 71 | 59 | 67 | 197
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5 | 10
  Asian | 3 | 1 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 15 | 13 | 13 | 41
  White | 48 | 50 | 44 | 142
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference Subscale of Brief Pain Inventory (BPI)
Description: The primary outcome is the Brief Pain Inventory Short Form Interference subscale (BPI). This is a 7-item scale that assesses the extent to which pain interferes with activities in daily life, such as general activity, mood, walking ability, work, relations with other people, sleep, and enjoyment of life. Scores range from 0 to 10 with higher scores indicating greater pain interference.
Time Frame: Baseline, Immediate post-treatment, 6 months after completing treatment
Population: Some participants did not complete the post-treatment and 6-month follow-up assessments. The main analyses that will be shared in publication are intent-to-treat but the means below reflect only those with complete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction (MBSR) | Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) | Usual Care
Number analyzed (Participants) | 75 | 71 | 71
score on a scale
  Baseline | 4.7 (2.2) | 4.8 (2.2) | 4.9 (2.2)
  Post-treatment: number analyzed (Participants) | 68 | 68 | 70
  Post-treatment | 4.4 (2.3) | 3.7 (2.0) | 4.8 (2.2)
  6-month follow-up: number analyzed (Participants) | 66 | 65 | 69
  6-month follow-up | 4.4 (2.6) | 3.8 (2.2) | 4.9 (2.5)

ADVERSE EVENTS:
Time Frame: 9 months (baseline to 6-months post-treatment assessment)
Description: Study definition conforms to clinicaltrials.gov definition
Arm/Group | Mindfulness-Based Stress Reduction (MBSR) | Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/75 | 1/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/75 | 0/71 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Stress Reduction (MBSR) (N=75) | Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) (N=71) | Usual Care (N=71)
Hospitalization (not study related) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (not study related) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04486066/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT04486066/ICF_002.pdf